CLINICAL TRIAL: NCT05829291
Title: A Feasibility and Safety Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Liver Metastases
Brief Title: Alpha Radiation Emitters Device for the Treatment of Liver Metastases (DaRT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-LIV-00
Record Dates: First submitted 2023-02-27; First posted 2023-04-25 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Liver Metastases
Keywords: Alpha radiation; Alpha emitting radiation; Liver Metastases; Brachytherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Diffusing Alpha Radiation Emitters Therapy (DaRT) — Alpha DaRT Applicators (the Alpha Needle Applicator, the Alpha Flex Applicator, and the Alpha Plant Applicator) and radioactive sources named Alpha DaRT Seeds - Ra-224 coated onto stainless steel tubes inserted into the tumor. Collectively, the Alpha DaRT Applicators and Seeds are referred to as the "Alpha DaRT Device".

SUMMARY:
This is a single center study enrolling up to 10 patients. The primary objective is to Evaluate the feasibility and safety of the DaRT for the treatment of Liver Metastases. The secondary objective is to evaluate the pathological response of liver metastases according to the Modified tumor regression grade[1] and to evaluate the radiological response of liver metastases using the RECIST criteria.

DETAILED DESCRIPTION:
This study is a Prospective, Open label, one arm, single center study to evaluate the feasibility and safety of Diffusing Alpha Radiation Emitters for the treatment of Liver Metastases .

Alpha Tau Medical proposes a unique treatment methodology for patients with liver metastases - Diffusing Alpha-emitters Radiation Therapy (DaRT) - whereby alpha particles are used to destroy solid tumors. The concept is predicated on the use of DaRT radioactive sources for radiotherapy.

DaRT is based on a nuclear decay chain originating with thorium-228 (1.91 years half-life). Outside of negligible, non-significant trace amounts, the thorium-228 remains confined to the Alpha Tau Medical manufacturing facility, and is used to generate radium-224, which is coated onto 316LVM stainless steel wires (Alpha DaRT Seeds).

The Primary endpoint of the study is : 1) Feasibility assessments of the ability to achieve full volume coverage of liver metastases volume.

2) Safety of the Alpha DaRT Seeds as therapy for liver metastases , Safety will be assessed and recorded according to CTCAE V5.

ELIGIBILITY:
Inclusion Criteria:

1. Referred for a two staged hepatectomy following a multidisciplinary team discussion, to resect liver metastases of colorectal cancer
2. Targetable lesion(s) must be technically amenable for complete coverage (including margins) by the Alpha DaRT Seeds / Target(s) must be reachable for implantation
3. Liver lesions are visible and measurable by CT according to RECIST v 1.1
4. Age ≥ 18 years old
5. ECOG Performance Status Scale ≤ 2
6. Subjects' life expectancy is at least 12 weeks
7. The following laboratory parameters

   * WBC ≥ 3500/µl, granulocyte ≥ 1500/µl
   * Hemoglobin > 85 g/L
   * Total bilirubin < 51.3 umol/L
   * Platelet count >75 X 109 /L or > 50% Prothrombin activity
   * Amylase and lipase < 1.5 X the upper limit of normal
   * AST and ALT ≤ 5 X ULN
   * Prothrombin time (PT) international normalized ratio (INR) < 2.3 or PT < 6 seconds above control. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists
8. Subjects are willing and able to sign an informed consent form
9. Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test within seven days before the Ra-224 implantation
10. Subjects must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy

Exclusion Criteria:

1. Concurrent cancer that is distinct in primary site or histology from colorectal cancer. Except cervical carcinoma in situ, prostate cancer with good prognosis, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated 3 years prior to entry is permitted.
2. Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids
3. Contraindication to angiography:

   * Any bleeding diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agent
   * Severe peripheral vascular disease precluding catheterization
   * History of severe allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically
4. Known hypersensitivity to any of the components of the treatment.
5. Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
6. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
7. Brain metastases
8. Active clinically serious infections
9. Major surgery within 4 weeks of start of the study therapy
10. Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
11. Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
12. High probability of protocol non-compliance (in opinion of investigator)
13. Pregnant or breastfeeding women
14. Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility - DaRT seed placement | From first operation - DaRT insertion up to 24 months
  Assessment of successful placement of the Alpha DaRT Seeds into liver metastases during a 2-stage hepatectomy via imaging
Safety - Adverse events | Up to 24 months
  Assess the frequency and severity of acute adverse events related to DaRT. Adverse events will be assessed and graded according to Common Terminology and Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
To evaluate the pathological response of liver metastases according to the Modified tumor regression grade 1 | 7-9 Weeks post DaRT insertion
  Pathological response to Alpha DaRT Seeds in covered areas after surgery
To evaluate the radiological response of liver metastases using the RECIST criteria . | 6-8 weeks post DaRT insertion
  Radiological response to Alpha DaRT seeds implantation after the Alpha DaRT Seeds insertion procedure and prior to the second stage

CONTACTS AND LOCATIONS:
Overall Officials: Peter Metrakos, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- e McGill University Health Centre (MUHC), Montreal, Quebec, Canada